CLINICAL TRIAL: NCT01852201
Title: POSITIVE: PerfusiOn Imaging Selection of Ischemic STroke PatIents for EndoVascular ThErapy
Brief Title: POSITIVE Stroke Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PRO23329
Record Dates: First submitted 2013-04-23; First posted 2013-05-13 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best medical therapy (No Intervention): Patients randomized to the control group will receive best conventional MT for acute ischemic stroke as determined by the attending stroke physician. Standardization of medical management in both arms will occur according to the following:
  * General medical management according to AHA/ASA guidelines
  * Admission to monitored or intensive care unit for at least 24 hours
  * Aggressive hypertensive-hypervolemic therapy should be used only in the case of symptomatic blood pressure fluctuations or if blood pressure drops below the normal range for the patient
  * Antithrombotics: ASA 325 mg PO qd for 7 days (clopidogrel may be used as adjunctive therapy if indicated for cardiac disease) then per discretion of treating physician
  * Close monitoring of BP and glucose with treatment according to AHA/ASA guidelines
  * Follow-up imaging study required in any patient with neurologic deterioration
- Endovascular treatment (Experimental): Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Interventions: Device: Endovascular Mechanical Thrombectomy

INTERVENTIONS:
Device: Endovascular Mechanical Thrombectomy — Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Other Names: mechanical revascularization
  Arms: Endovascular treatment

SUMMARY:
Primary Endpoint:

The primary objective is to show that AIS patients, ineligible for or refractory to treatment with IV-tPA, with appropriate image selection, treated with mechanical thrombectomy within 6-12 hours of symptom onset have less stroke related disability and improved good functional outcomes as compared to those treated with best MT with respect to endpoint defined as:

• 90-day global disability assessed via the modified Rankin score (mRS), analyzed using raw mRS scores. Statistical details can be found in section 7.2.

Secondary Endpoints:

* 90-day global disability in the 6-12 hr cohort assessed via the overall distribution of mRS
* Proportion of patients with good functional recovery for the 6-12 hr cohort as defined by mRS 0-2 at 90 days
* Mortality at 30 and 90 days
* Intracranial hemorrhage with neurological deterioration (NIHSS worsening >4) within 24 hours of randomization
* Procedure related serious adverse events (SAE's)
* Arterial revascularization measured by TICI 2b or 3 following device use

DETAILED DESCRIPTION:
Intravenous (IV) tissue plasminogen activator (tPA) administration has been shown to be safe and effective for treatment of AIS within 3 hours of symptom onset, and newer evidence has shown potential benefit out to 4.5 hours. Mechanical thrombectomy for AIS patients has been shown in clinical trials to be safe up to 8 hours after symptom onset. The rapid progression of thrombectomy devices over the last several years has resulted in faster recanalization times while maintaining a high degree of safety. This has resulted in improved patient outcomes, similar to prior randomized trial data showing improved outcomes over medical therapy or earlier devices. Data from the MERCI trial suggests that patients > 85 as well as those with a baseline NIHSS score > 30 are unlikely to benefit from thrombectomy. Patients with rapidly improving neurologic deficits likely will have an excellent recovery with conventional care, precluding the ability to detect a beneficial treatment effect of thrombectomy.

Pilot data incorporating physiologic imaging has shown that appropriate patients can be selected for thrombectomy. This selection methodology has shown the ability to maintain the same level of safety and efficacy as those patients treated in the highly selective environment of a clinical trial, despite presenting far beyond accepted time based standards. Vertebrobasilar occlusion patients are excluded to maintain a homogenous study population, particularly since no data currently is available addressing the comparability of imaging penumbral patterns in the anterior vs. posterior circulation. This has also been shown to be reproducible at multiple centers and with different imaging modalities. However, all prospective interventional stroke studies performed to date have been restricted by the 8-hour time window.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older (i.e., candidates must have had their 18th birthday)
2. NIHSS ≥8 at the time of neuroimaging
3. Presenting or persistent symptoms within 6-12 hours of when groin puncture can be obtained
4. Neuroimaging demonstrates large vessel proximal occlusion (distal ICA through MCA M1 bifurcation)
5. The operator feels that the stroke can be appropriately treated with traditional endovascular techniques (endovascular mechanical thrombectomy without adjunctive devices such as stents)
6. Pts are within 6-12 hours of symptom onset, that have received IV-tPA without improvement in symptoms are eligible for this study. Patients presenting earlier than 6 hours should be treated according to local standard of care.
7. Pre-event Modified Rankin Scale score 0-1
8. Consenting requirements met according to local IRB

Exclusion Criteria:

1. Patient is less than 6-hours from symptom onset
2. Rapidly improving neurologic examination
3. Absence of large vessel occlusion on non-invasive imaging
4. Known or suspected pre-existing (chronic) large vessel occlusion in the symptomatic territory
5. Absence of an associated large penumbra as defined by physiologic imaging according to standard of practice at the participating institution
6. Any intracranial hemorrhage in the last 90 days
7. Known irreversible bleeding disorder
8. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 2.5 or institutionally equivalent prothrombin time of 2.5 times normal
9. Platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
10. Inability to tolerate, clinically documented evidence in medical history of adverse reaction to, or contraindication to medications used in treatment of the stroke
11. Contraindication to CT and MRI (i.e., iodine contrast allergy or other condition that prohibits imaging from either CT or MRI)
12. Known allergy to contrast used in angiography that cannot be medically controlled
13. Relative contraindication to angiography (e.g., serum creatinine > 2.5 mg/dL)
14. Women who are currently pregnant or breast-feeding (Women of child-bearing potential must have a negative pregnancy test prior to the study procedure (either serum or urine)
15. Evidence of active infection (indicated by fever at or over 99.9 °F and/or open draining wound) at the time of randomization
16. Current use of cocaine or other vasoactive substance
17. Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 90 days
18. Patients who lack the necessary mental capacity to participate or are unwilling or unable to comply with the protocol's follow up appointment schedule (based on the investigator's judgment)

Head CT or MRI Scan Exclusion Criteria

* Presence of blood on imaging (subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH), etc.)
* High density lesion consistent with hemorrhage of any degree
* Significant mass effect with midline shift
* Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan or ASPECTS of < 7; Sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lena, MD, Principal Investigator — Medical University of South Carolina
Locations (20):
- United States (20):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Swedish/Colorado Neurological Institute, Englewood, Colorado
  - Baptist Health, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Univesity of Massachusetts-Worcester, Worcester, Massachusetts
  - Saint Luke's Hospital, Kansas City, Missouri
  - Captial Health, Trenton, New Jersey
  - University of Buffalo Neurosurgery, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Stony Brook Medical Center, Stony Brook, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Interventional Associates, Chattanooga, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist Healthcare - Memphis, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - West Virginia University, Morgantown, West Virginia
  - Wisconsin University, Madison, Wisconsin

REFERENCES:
- [Derived] Roaldsen MB, Jusufovic M, Berge E, Lindekleiv H. Endovascular thrombectomy and intra-arterial interventions for acute ischaemic stroke. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD007574. doi: 10.1002/14651858.CD007574.pub3. PMID 34125952
- [Derived] Mocco J, Siddiqui AH, Fiorella D, Alexander MJ, Arthur AS, Baxter BW, Budzik RF, Froehler MT, Hanel RA, Lena J, Persaud S, Puri AS, Rai AT, Wintermark M, Woodward K, Zhang X, Turk A. POSITIVE: Perfusion imaging selection of ischemic stroke patients for endovascular therapy. J Neurointerv Surg. 2022 Feb;14(2):126-132. doi: 10.1136/neurintsurg-2021-017315. Epub 2021 Feb 25. PMID 33632884

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Therapy: Patients randomized to the control group will receive best conventional MT for acute ischemic stroke as determined by the attending stroke physician. Standardization of medical management in both arms will occur according to the following:
  * General medical management according to AHA/ASA guidelines
  * Admission to monitored or intensive care unit for at least 24 hours
  * Aggressive hypertensive-hypervolemic therapy should be used only in the case of symptomatic blood pressure fluctuations or if blood pressure drops below the normal range for the patient
  * Antithrombotics: ASA 325 mg PO qd for 7 days (clopidogrel may be used as adjunctive therapy if indicated for cardiac disease) then per discretion of treating physician
  * Close monitoring of BP and glucose with treatment according to AHA/ASA guidelines
  * Follow-up imaging study required in any patient with neurologic deterioration
- Endovascular Treatment (Thrombectomy Procedure: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Endovascular Mechanical Thrombectomy: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical r
Period: Overall Study
Arm/Group | Medical Therapy | Endovascular Treatment (Thrombectomy Procedure
Started | 21 | 12
Completed | 21 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Endovascular Treatment: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Endovascular Mechanical Thrombectomy: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical r
- Total: Total of all reporting groups
Arm/Group | Best Medical Therapy | Endovascular Treatment | Total
Number analyzed (Participants) | 21 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13) | 70 (10.1) | 67 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 12 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: Rate of Good Functional Outcomes Measured by Modified Rankin Score (mRS)
Description: Modified rankin score measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The range is 0-6 (0 is highest function with no symptoms and 6 is death). This outcome measured percentage of subjects with a "good" functional outcome with a score ranging from 0-2.
  The primary objective is to show that AIS patients, ineligible for or refractory to treatment with IV-tPA, (patients seen within 6 hours of symptom onset will be immediately considered for endovascular therapy according to the site's standard of care. Likewise, patients presenting beyond 12 hours will be treated according to the site's standard of care), with appropriate image selection, treated with mechanical thrombectomy within 6-12 hours of symptom onset have less stroke related disability and improved good functional outcomes as compared to those treated with best MT.
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Groups:
- Endovascular Treatment: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Endovascular Mechanical Thrombectomy: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revas
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 21 | 12
percentage of participants | 42.9 | 75

2. Secondary Outcome: Percentage of Participants in the 6-12 hr Cohort With Global Disability as Assessed by the Modified Rankin Score (mRS)
Description: The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. A score of 3-6 represents global disability are defined as follows: (3) moderate disability (requiring some help, but able to walk without assistance); (4) moderate severe disability (unable to walk without assistance and unable to attend to own bodily needs without assistance); (5) severe disability (bedridden, incontinent and requiring constant nursing care and attention; and (6) dead.
Time Frame: 90 day
Population: There were only 12 participants total in the 6-12hr cohort
Measure: Number; unit: percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 8 | 4
percentage of participants | 62.5 | 50

3. Secondary Outcome: Percentage of Participants in the 6-12hr Cohort With Good Functional Recovery as Assessed by the Modified Rankin Scale (mRS)
Description: The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. A score of 0-2 represents good functional recovery. The scores are defined as follows: (0) No symptoms at all; (1) No significant disability despite symptoms, able to carry out all usual duties and activities; (2) Slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance.
Time Frame: 90 days
Measure: Number; unit: Percentage of particpants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 21 | 12
Percentage of particpants | 42.9 | 75.0

4. Secondary Outcome: Percentage of Participants Mortality at 30 Days
Description: Mortality at 30 days will be compared between randomized groups in an ITT fashion; with overall Type I error controlled using hierarchical testing. That is, if statistical significance is observed on the primary effectiveness endpoint, the secondary clinical efficacy endpoints will then be tested in sequential fashion each at a two-sided alpha level of 0.05, with testing ceasing once a null hypothesis cannot be rejected.
Time Frame: 30 days
Population: The values for 4 subjects was not captured at this timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 17 | 12
percentage of participants | 12 | 0

5. Secondary Outcome: Percentage of Participants Mortality at 90 Days
Description: Mortality at 90 days will be compared between randomized groups in an ITT fashion; with overall Type I error controlled using hierarchical testing. That is, if statistical significance is observed on the primary effectiveness endpoint, the secondary clinical efficacy endpoints will then be tested in sequential fashion each at a two-sided alpha level of 0.05, with testing ceasing once a null hypothesis cannot be rejected.
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 21 | 12
percentage of participants | 19.1 | 8.3

6. Secondary Outcome: Percentage of Participants With ICH (Intracranial Hemorrhage) With Neurological Deterioration (NIHSS Worsening >4).
Description: ICH with neurological deterioration (NIHSS worsening >4) will be compared between randomized groups in an ITT fashion; with overall Type I error controlled using hierarchical testing. That is, if statistical significance is observed on the primary effectiveness endpoint, the secondary clinical efficacy endpoints will then be tested in sequential fashion each at a two-sided alpha level of 0.05, with testing ceasing once a null hypothesis cannot be rejected.
Time Frame: 90 days
Population: One patient had no NIHSS scores after baseline and was excluded from this analysis
Measure: Number; unit: percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 20 | 12
percentage of participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With SAE's Related to a Thrombectomy Procedure
Description: A Thrombectomy is an interventional procedure to remove a blood clot (thrombus) from a blood vessel in the brain.
  Procedure related SAE's will be compared between randomized groups in an ITT fashion; with overall Type I error controlled using hierarchical testing. That is, if statistical significance is observed on the primary effectiveness endpoint, the secondary clinical efficacy endpoints will then be tested in sequential fashion each at a two-sided alpha level of 0.05, with testing ceasing once a null hypothesis cannot be rejected.
Time Frame: 90 days
Measure: Number; unit: Percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 21 | 12
Percentage of participants | 0.0 | 8.3

8. Secondary Outcome: Arterial Revascularization Measured by TICI 2b or 3 Following Device Use
Description: Arterial revascularization measured by TICI 2b or 3 following device use will be compared between randomized groups in an ITT fashion; with overall Type I error controlled using hierarchical testing. That is, if statistical significance is observed on the primary effectiveness endpoint, the secondary clinical efficacy endpoints will then be tested in sequential fashion each at a two-sided alpha level of 0.05, with testing ceasing once a null hypothesis cannot be rejected.
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 1 | 12
percentage of participants | 100 | 83

9. Secondary Outcome: Percentage of Patients With Serious Adverse Events (SAEs) Related to Thrombectomy Device.
Description: A Thrombectomy device is a device intended to restore blood flow in a vessel in the brain by removing a blood clot (thrombus).
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Arm/Group | Best Medical Therapy | Endovascular Treatment
Number analyzed (Participants) | 21 | 12
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study-104 days
Groups:
- Endovascular Treatment: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Endovascular Mechanical Thrombectomy: Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical re
Arm/Group | Best Medical Therapy | Endovascular Treatment
All-Cause Mortality (participants affected / at risk) | 4/21 | 1/12
Serious Adverse Events (participants affected / at risk) | 12/21 | 4/12
Other Adverse Events (participants affected / at risk) | 10/21 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Best Medical Therapy (N=21) | Endovascular Treatment (N=12)
Asymptomatic intracranial hemorrhage up to 24 hours post-randomization (Vascular disorders) | 2 (2) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheal thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Worsening of pre-exist. cond.- Severely reduced LV, mildly reduced RV systolic function (Vascular disorders) | 1 (1) | 0 (0)
Neurologic Deterioration (Vascular disorders) | 3 (4) | 0 (0)
Emboli (Vascular disorders) | 1 (1) | 0 (0)
Myocardioal Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Infected PICC Line (Infections and infestations) | 1 (1) | 0 (0)
Worsening of Pre Existing Condition-Mid Sternal Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Worsening of Pre Existing Condition-Diffuse encephalopathy and cortical irritability (Vascular disorders) | 1 (1) | 0 (0)
dysphasia (Vascular disorders) | 1 (1) | 0 (0)
Worsening of Index Stroke (Vascular disorders) | 1 (1) | 0 (0)
Pneumothorax (Vascular disorders) | 1 (1) | 0 (0)
Inability to Feed (Gastrointestinal disorders) | 1 (1) | 0 (0)
L Hip dislocation requiring closed reduction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Troponinemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Metabolic Encephalopathy (Vascular disorders) | 1 (1) | 0 (0)
Altered Mental Status (General disorders) | 1 (1) | 0 (0)
Febrile with Chest Pain (General disorders) | 1 (1) | 0 (0)
Failure to thrive (General disorders) | 1 (1) | 0 (0)
Accidental narcotic overdose (General disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Best Medical Therapy (N=21) | Endovascular Treatment (N=12)
Groin puncture site: hematoma (Vascular disorders) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 2 (2) | 1 (1)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Distal Emboli (Vascular disorders) | 0 (0) | 2 (2)
Neurological Deterioration (increase of >4 points on NIHSS) (Vascular disorders) | 3 (3) | 0 (0)
Bactermia (Infections and infestations) | 2 (2) | 0 (0)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hemorrhagic Conversion (Vascular disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT01852201/Prot_SAP_000.pdf